CLINICAL TRIAL: NCT02688803
Title: Multicentre Study to Determine the Feasibility of Using an Integrated Consent Model to Compare Three Standard of Care Regimens for The Treatment of Triple-Negative Breast Cancer in the Neoadjuvant/Adjuvant Setting (REaCT-TNBC) OTT 15-04
Brief Title: Multicentre Study to Determine the Feasibility of Using an Integrated Consent Model to Compare Three Standard of Care Regimens for The Treatment of Triple-Negative Breast Cancer in the Neoadjuvant/Adjuvant Setting (REaCT-TNBC)
Acronym: OTT15-04
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study did not meet the pilot feasibility endpoints and was formally closed to accrual prematurely on February 8, 2017.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20160078-01H
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: HER2 Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Fluorouracil; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose dense AC-P (Active Comparator): Dose dense AC-P (doxorubicin 60 mg/m2 plus cyclophosphamide 600 mg/m2 q2weeks x 4 cycles followed by paclitaxel 175 mg/m2 q2weeks x 4 cycles)
  Interventions: Drug: Dose dense AC-P
- Dose dense AC (Active Comparator): Dose dense AC followed by weekly P (doxorubicin 60 mg/m2 plus cyclophosphamide 600 mg/m2 q2weeks x 4 cycles followed by paclitaxel 80 mg/m2 weekly x 12 cycles)
  Interventions: Drug: Dose dense AC
- FEC-D (Active Comparator): FEC-D (5-FU 500 mg/m2 plus epirubicin 100 mg/m2 plus cyclophosphamide 500 mg/m2 q3weeks x 3 cycles followed by docetaxel 100 mg/m2 q3weeks x 3 cycles)
  Interventions: Drug: FEC-D

INTERVENTIONS:
Drug: Dose dense AC-P — (doxorubicin 60 mg/m2 plus cyclophosphamide 600 mg/m2 q2weeks x 4 cycles followed by paclitaxel 175 mg/m2 q2weeks x 4 cycles)
  Other Names: doxorubicin; cyclophosphamide; paclitaxel
  Arms: Dose dense AC-P
Drug: Dose dense AC — Dose dense AC followed by weekly P (doxorubicin 60 mg/m2 plus cyclophosphamide 600 mg/m2 q2weeks x 4 cycles followed by paclitaxel 80 mg/m2 weekly x 12 cycles)
  Other Names: doxorubicin; cyclophosphamide; paclitaxel
  Arms: Dose dense AC
Drug: FEC-D — FEC-D (5-FU 500 mg/m2 plus epirubicin 100 mg/m2 plus cyclophosphamide 500 mg/m2 q3weeks x 3 cycles followed by docetaxel 100 mg/m2 q3weeks x 3 cycles)
  Other Names: 5-FU; cyclophosphamide; docetaxel
  Arms: FEC-D

SUMMARY:
Triple-negative breast cancer (TNBC) is a term applied to breast cancer cases that have <1% expression of the estrogen receptor (ER) and the progesterone receptor (PR) and do not over express HER2.

TNBC is diagnosed in 15-20% of breast cancer cases and tends to occur in younger women and have biologically more aggressive high grade disease. Clinically, patients with TNBC have a poorer prognosis compared to patients diagnosed with other breast cancer subtypes. Because of the aggressive phenotype and due to observations that systemic chemotherapy offers significantly higher benefit in ER negative disease, current treatment guidelines from provincial and other organizations recommend that patients receive adjuvant systemic chemotherapy for any TNBC greater than 0.5 cm in greatest diameter or node positive independent of primary tumor size.

Currently, there is no world-wide standard recommended chemotherapy regimen for the management of TNBC in the neoadjuvant/adjuvant setting, with treatments varying from region and institution.

As physicians do not know what the "best" treatment for patients is, genuine uncertainty ("clinical equipoise") exists. Physicians will choose between different "standards" in their personal practice, using idiosyncratic decision making processes, without the physician or the patient knowing the optimal option. This is not good for patients, physicians and society as a whole. Determining the optimal treatment remains an important medical issue for patients, physicians and society. This study will survey opinions on a novel method to allow comparisons of established standard of care prophylactic treatment using the "integrated consent model" as part of a pragmatic clinical trial and attempt to compare head to head standard chemotherapy regimens in patients with TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary TNBC breast cancer
* Planned for chemotherapy
* ≥18 years of age
* Able to provide verbal consent
* Willing to complete a survey

Exclusion Criteria:

* Metastatic disease
* Contraindication to one or more of the chemotherapy agents being evaluated in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hilton, Dr., Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobs C, Clemons M, Mazzarello S, Hutton B, Joy AA, Brackstone M, Freedman O, Vandermeer L, Ibrahim M, Fergusson D, Hilton J. Enhancing accrual to chemotherapy trials for patients with early stage triple-negative breast cancer: a survey of physicians and patients. Support Care Cancer. 2017 Jun;25(6):1881-1886. doi: 10.1007/s00520-017-3580-4. Epub 2017 Jan 27. PMID 28127659
- [Result] Hilton J, Stober C, Mazzarello S, Vandermeer L, Fergusson D, Hutton B, Clemons M. Randomised feasibility trial to compare three standard of care chemotherapy regimens for early stage triple-negative breast cancer (REaCT-TNBC trial). PLoS One. 2018 Jul 24;13(7):e0199297. doi: 10.1371/journal.pone.0199297. eCollection 2018. PMID 30040817
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/studies/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 patients were approached for the study between August 30, 2016 and January 31, 2017, and both were enrolled and randomized. The study was closed to accrual prematurely on February 8, 2017, because it did not meet the pilot feasibility endpoints. According to the protocol, feasibility success is defined as over 50% of appropriate patients approached agree to participate, and over 50% of physicians who agree to participate approached patients for the study.
Period: Overall Study
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Started | 1 | 0 | 1
Completed | 1 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the Dose Dense AC group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D | Total
Number analyzed (Participants) | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected. This was a feasibility study.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex variable was not collected. This was a feasibility study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 1 |  | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Receive Chemotherapy in the Neoadjuvant/Adjuvant Setting for TNBC
Description: Percentage of patients who receive chemotherapy in the neoadjuvant/adjuvant setting for TNBC compared to the number of participants who after being approached subsequently agree to randomization.
Time Frame: One year
Population: 2 patients were approached for the study and randomized. The study did not meet feasibility and accrual was closed early.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Number analyzed (Participants) | 1 | 0 | 1
Participants
  Received chemotherapy | 1 |  | 1
  Chemotherapy dose adjustments or delays | 0 |  | 1
  Completed study as planned | 0 |  | 1

2. Primary Outcome: Participant Satisfaction
Description: Participant satisfaction survey. Overall participant satisfaction will be determined using the participant survey
Time Frame: One year
Population: No participants were randomized to the Dose-dense AC group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Number analyzed (Participants) | 1 | 0 | 1
Participants
  The clinical trial was explained clearly to me by my oncologist.: Strongly disagree | 0 |  | 0
  The clinical trial was explained clearly to me by my oncologist.: Disagree | 0 |  | 0
  The clinical trial was explained clearly to me by my oncologist.: Neutral | 0 |  | 0
  The clinical trial was explained clearly to me by my oncologist.: Agree | 1 |  | 1
  The clinical trial was explained clearly to me by my oncologist.: Strongly agree | 0 |  | 0
  The clinical trial was explained clearly to me by my oncologist.: Not applicable | 0 |  | 0
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Strongly disagree | 0 |  | 0
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Disagree | 0 |  | 0
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Neutral | 0 |  | 0
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Agree | 1 |  | 1
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Strongly agree | 0 |  | 0
  I thought that the questions I had about the clinical trial were answered to my satisfaction.: Not applicable | 0 |  | 0
  If I was asked to participate in this study again, I would say yes.: Strongly disagree | 0 |  | 0
  If I was asked to participate in this study again, I would say yes.: Disagree | 0 |  | 0
  If I was asked to participate in this study again, I would say yes.: Neutral | 0 |  | 0
  If I was asked to participate in this study again, I would say yes.: Agree | 1 |  | 1
  If I was asked to participate in this study again, I would say yes.: Strongly agree | 0 |  | 0
  If I was asked to participate in this study again, I would say yes.: Not applicable | 0 |  | 0
  I found that taking part in this study interfered with my quality of life.: Strongly disagree | 0 |  | 0
  I found that taking part in this study interfered with my quality of life.: Disagree | 1 |  | 1
  I found that taking part in this study interfered with my quality of life.: Neutral | 0 |  | 0
  I found that taking part in this study interfered with my quality of life.: Agree | 0 |  | 0
  I found that taking part in this study interfered with my quality of life.: Strongly agree | 0 |  | 0
  I found that taking part in this study interfered with my quality of life.: Not applicable | 0 |  | 0
  I found that it was time-consuming to take part in this study.: Strongly disagree | 0 |  | 0
  I found that it was time-consuming to take part in this study.: Disagree | 1 |  | 1
  I found that it was time-consuming to take part in this study.: Neutral | 0 |  | 0
  I found that it was time-consuming to take part in this study.: Agree | 0 |  | 0
  I found that it was time-consuming to take part in this study.: Strongly agree | 0 |  | 0
  I found that it was time-consuming to take part in this study.: Not applicable | 0 |  | 0

3. Secondary Outcome: Percentage of Participants Who Complete Study Treatment
Description: Percentage of participants who complete study treatment compared to the percentage who discontinue their treatment while on study (compliance) will be calculated using the sites chemotherapy treatment records and data from New Patient Registration.
Time Frame: One year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Number analyzed (Participants) | 1 | 0 | 1
Participants | 0 | 0 | 1

4. Secondary Outcome: Hospitalization
Description: The number of participants with adverse effects requiring hospitalization
Time Frame: One year
Population: There were no participants randomized to the Dose Dense AC group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Number analyzed (Participants) | 1 | 0 | 1
Participants | 0 |  | 0

5. Secondary Outcome: Treatment Delays
Description: The number of participants with adverse effects requiring treatment delays
Time Frame: One year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
Number analyzed (Participants) | 1 | 0 | 1
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was followed for approximately one year.
Description: Serious Adverse Event (SAE) reporting is not required for this feasibility study, as per the protocol. Adverse events were not collected or reported. Secondary outcomes of hospitalization/treatment delays were collected by a variety of study staff on the case report forms, however they were not graded as adverse events. As per the protocol, there were no additional risks associated with this study as all arms are standard of care in this pragmatic clinical trial.
Arm/Group | Dose Dense AC-P | Dose Dense AC | FEC-D
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study did not meet feasibility and was terminated early. The study only involved 2 cancer centres. Physicians reported few TNBC patients in their clinics, and that it was challenging to tell a TNBC patient that the optimal chemotherapy regimen for their condition is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT02688803/Prot_SAP_000.pdf